The Effect of Music Integrated Phonological Awareness Program on Phonological Awareness Skills of Preschool (5-6 Years) Cochlear Implant Users

## **Informed Consent Form**

This study you participated in is a scientific research and the name of the research is "The Effect of Music Integration Phonological Awareness Program on Preschool Cochlear Implant Users".

The study will be carried out within the body of Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Department of Otorhinolaryngology, Hearing and Speech Disorders, and as an institution, the necessary personnel and equipment infrastructure are available to continue these studies.

It is expected that 46 participants will participate in our research. It is planned that all measurements and evaluations for each participant will be completed within an estimated 1 hour.

Procedures to be applied:

The procedures to be performed do not include any medical intervention.

The measurements to be made to the candidates within the scope of this study do not contain any harmful effects. First, the patient who will undergo a spectral modulated ripple test (SMRT) will be asked to say the different sound he/she hears. Then the auditory system will be evaluated in auditory evoked late potentials (AIP). Afterwards, the phonological awareness level will be determined by the phonological awareness test.

No treatment procedure or alternative treatment methods will be applied in the study.

Risks:

There is no application and risk that will affect the health integrity of the person.

Participant Rights and Responsibilities:

All data obtained will be stored in accordance with the privacy policy. The data to be obtained will not be made public. In the data to be used in the study, the names of the individuals will be kept confidential.

When there is a change in the research or research method, this will be communicated to the participants or their legal representatives in a timely manner and they will be informed.

Measurement results and personal information will not be shared in any environment, and will only be given to you if you request it.

In the transactions to be made; You will not be charged any fees. You will not be charged any fees. No fee will be charged from the Social Security Institution (SGK) to which you are affiliated.

Participation in the study is on a voluntary basis. As a participant, you can refuse to participate in the research or withdraw from the research at any time, with or without justification, without incurring any penalty or sanction, without losing any of your rights.

As a participant during the study, it is his responsibility to carefully follow the instructions given by the person conducting the study.

**Volunteering Statement:** 

The research in question; Since it was clearly explained to me that I could participate in my own free will without any coercion, that I could leave the study group whenever I wanted, that if I participated, no fee would be charged to me or the institution, that my personal information would not be shared in any medium, that these tests would not have any harmful effects, and that I could join this study group. I accept as I don't mind participating.

I have read all the explanations in the Informed Consent Form. Written and verbal explanations regarding the research, the subject and purpose of which are stated above, were given to me by the expert named below. I know that I have voluntarily participated in the research and will leave the research at any time, with or without justification.

Participant Name and Surname: Explanatory Name and Surname:

Ody. Büşra YILANLI

**Date:** 08.03.2021 **Date:** 08.03.2021

Phone number: Phone Number: 0535 261 1050

Sign: Sign: